CLINICAL TRIAL: NCT05760924
Title: Randomized Trial of Left Bundle Branch Pacing Effect on Clinical Outcomes and Left Ventricular Remodeling in Patients With Nonresponse to Biventricular Cardiac Resynchronization Therapy
Brief Title: Left Bundle Branch Pacing on Outcomes and Ventricular Remodeling in Biventricular CRT Nonresponders
Acronym: RESCUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Tariel A. Atabekov, Medical Doctor, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE
Record Dates: First submitted 2023-02-22; First posted 2023-03-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Left Bundle-Branch Block; Ischemic Cardiomyopathy; Non-ischemic Dilated Cardiomyopathy; Left Ventricular Dysfunction; Left Ventricle Remodeling
Keywords: Cardiac Resynchronization Therapy; Biventricular Pacing; Left Bundle Branch Pacing; Speckle Tracking Echocardiography; Biomarker of Fibrosis and Remodeling; Combined Left Bundle Branch and Left Ventricular Pacing; CRT Non-responder; CRT Responder
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block; Ventricular Dysfunction, Left; Ventricular Remodeling | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cardiac Resynchronization Therapy with Biventricular Pacing (Active Comparator): Patients who are non-responders to biventricular cardiac resynchronization therapy (CRT) with indications to CRT devices with defibrillator function (CRT-D) or CRT-D leads replacement. CRT-D or CRT-D leads replacement will be performed in this group of patients.
  Interventions: Device: Cardiac Resynchronization Therapy Devices with Defibrillator Function (CRT-D) or CRT-D Leads Replacement
- Cardiac Resynchronization Therapy with Left Bundle Branch Pacing (Experimental): Patients who are non-responders to biventricular cardiac resynchronization therapy (CRT) with indications to CRT devices with defibrillator function (CRT-D) or CRT-D leads replacement. CRT-D or CRT-D leads replacement with the new lead implantation to the left bundle branch and inactivation of conventional right and left ventricular pacing will be performed in this group of patients.
  Interventions: Device: CRT-D or CRT-D Leads Replacement with New Lead Implantation to Left Bundle Branch and Inactivation of Conventional Right and Left Ventricular Pacing
- Cardiac Resynchronization Therapy with Combined Left Bundle Branch and Left Ventricular Pacing (Experimental): Patients who are non-responders to biventricular cardiac resynchronization therapy (CRT) with indications to CRT devices with defibrillator function (CRT-D) or CRT-D leads replacement. CRT-D or CRT-D leads replacement with the new lead implantation to the left bundle branch and inactivation of conventional right ventricular pacing will be performed in this group of patients.
  Interventions: Device: CRT-D or CRT-D Leads Replacement with New Lead Implantation to Left Bundle Branch and Inactivation of Conventional Right Ventricular Pacing

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy Devices with Defibrillator Function (CRT-D) or CRT-D Leads Replacement — The local anesthesia will be performed on the left/right subclavian area after prepping the skin. The device pocket will be opened, the old CRT-D will be removed and disconnected from the leads. The pacing threshold, intracardiac signal amplitude and impedance (pacing and shock) on the atrial, defibrillation and left ventricular leads will be performed. If there is a lead dysfunction, the new lead will be implanted. The new CRT-D will be connected with leads and placed back into the pocket. The pocket will be closed by separate stitches (2-4 suffice) using the resorbable braided suture.
  Arms: Cardiac Resynchronization Therapy with Biventricular Pacing
Device: CRT-D or CRT-D Leads Replacement with New Lead Implantation to Left Bundle Branch and Inactivation of Conventional Right and Left Ventricular Pacing — The local anesthesia will be performed on the left/right subclavian area after prepping the skin. The device pocket will be opened, the old CRT-D will be removed and disconnected from the leads. The pacing threshold, intracardiac signal amplitude and impedance (pacing and shock) on the atrial, defibrillation and left ventricular leads will be performed. If there is a lead dysfunction, the new lead will be implanted. The lead implantation to the left bundle branch (LBB) will be performed by transvenous approach and special delivery system. The new CRT-D will be connected with the leads (LBB pacing lead will be connected to defibrillation lead (DL) IS-1 connector of CRT-D and IS-1 tip of DL will be capped) and placed back into pocket. The pocket will be closed by separate stitches (2-4 suffice) using the resorbable braided suture. RV and LV pacing will be inactivated and only LBB pacing will be switched on.
  Arms: Cardiac Resynchronization Therapy with Left Bundle Branch Pacing
Device: CRT-D or CRT-D Leads Replacement with New Lead Implantation to Left Bundle Branch and Inactivation of Conventional Right Ventricular Pacing — The local anesthesia will be performed on the left/right subclavian area after prepping the skin. The device pocket will be opened, the old CRT-D will be removed and disconnected from the leads. The pacing threshold, intracardiac signal amplitude and impedance (pacing and shock) on the atrial, defibrillation and left ventricular leads will be performed. If there is a lead dysfunction, the new lead will be implanted. The lead implantation to the left bundle branch (LBB) will be performed by transvenous approach and special delivery system. The new CRT-D will be connected with the leads (LBB pacing lead will be connected to defibrillation lead (DL) IS-1 connector of CRT-D and IS-1 tip of DL will be capped) and placed back into pocket. The pocket will be closed by separate stitches (2-4 suffice) using the resorbable braided suture. LBB and LV pacing will be switched on.
  Arms: Cardiac Resynchronization Therapy with Combined Left Bundle Branch and Left Ventricular Pacing

SUMMARY:
Heart failure (HF) is the most common nosology encountered in clinical practice. Its incidence and prevalence increase exponentially with increasing age and it is associated with the increased mortality, more frequent hospitalization and decreased quality of life. An initial approach to the treatment of HF patients with reduced left ventricular (LV) systolic function and left bundle branch block (LBBB) was implantation of device for cardiac resynchronization therapy using biventricular pacing. This has resulted in long-term clinical benefits such as improved quality of life, increased functional capacity, reduced HF hospitalizations and overall mortality. However, conventional cardiac resynchronization therapy (CRT) is effective in only 70% of patients. And the remaining 30% of patients are non-responders to conventional CRT. Cardiac conduction system pacing is currently a promising technique for these patients. Particularly, His bundle pacing (HBP) has been developed to achieve the same results. According to other studies HBP has shown greater improvement in hemodynamic parameters comparing with conventional biventricular CRT. But, nevertheless, there are significant clinical troubles with HBP, especially high pacing threshold. In this regard, in 2017, the left bundle branch pacing (LBBP) was developed, which demonstrated clinical advantages compared to conventional biventricular CRT. Also, since 2019, left bundle branch pacing-optimized CRT (LBBPO CRT) has been used in clinical practice. These methods have become an alternative to HBP due to the stimulation of LBB outside the blocking site, a stable pacing threshold and a narrow QRS complex duration on electrocardiogram. A series of case reports and observational studies have demonstrated the efficacy and safety of LBBP and LBBPO CRT in patients with CRT indications. However, it is not enough data about impact of CRT with LBBP and combined CRT with LBBP and LV pacing on myocardial remodeling, reducing mortality and complications. According to our hypothesis, CRT with LBBP and combined CRT with LBBP and LV pacing compared with conventional biventricular pacing will significantly improve the clinical outcomes and reverse myocardial remodeling in patients who are non-responders to biventricular CRT with HF, reduced LV ejection fraction and with indications to CRT devices with defibrillator function (CRT-D) or one of the CRT-D leads replacement.

DETAILED DESCRIPTION:
Recent advances in the cardiovascular pharmacological and cardiac device-based therapy have led to many benefits which improve the clinical condition, reduce morbidity, and increase survival in patients with heart failure (HF). Cardiac resynchronization therapy (CRT) with biventricular pacing is a well-established method for the treatment of patients with the left bundle branch block (LBBB), cardiomyopathy of difference etiologies and HF with the reduced left ventricular ejection fraction (LVEF). Several prospective randomized trials have shown that biventricular CRT improves quality of life, improves exercise tolerance, reduces HF hospitalizations, and reduces all-cause mortality. The enthusiasm for this remarkable efficacy of CRT is limited by the fact that a proportion of patients have no benefits from this treatment. This category of patients is called nonresponder. These patients have no clinical and echocardiographic improvement with CRT. According to some studies, 30-50% of patients with biventricular CRT are non-responders.

The left bundle branch pacing (LBBP) was proposed in 2017 and demonstrated clinical benefits in patients with HF and LBBB, aiming to pace the proximal left bundle branch (LBB) along with LV myocardial capture. During selective pacing, only LBB is captured without the nearby myocardium, while with non-selective LBBP the septal myocardium is captured. LBBP with lead implanted slightly distal to the His bundle and screwed deep into the left ventricular (LV) septum is ideal for LBB capture. LBBP has emerged as an alternative to HBP due to pacing outside the blocking site, a stable pacing threshold, and a narrow QRS complex duration on electrocardiogram in patients with the bradycardia. In some clinical cases for the first time was demonstrated that LBBP could lead to complete correction of LBBB and improvement in cardiac function in patients with LBBB and HF. In another observational study it was shown that LBBP could be a new method of CRT. Subsequently, several case reports and observational studies have demonstrated the efficacy and safety of LBBP in patients with indications for CRT device implantation.

However, proximal LBBP is inherently limited in its ability to restore the physiological activation of LV lateral wall in patients with the conduction delay in the distal segment of LBB, Purkinje fibers or LV myocardium. Moreover, it is possible that in many patients with LBBP, only LV septal myocardial capture has been obtained, resulting in a small but potentially important non-physiological delay in LV lateral wall activation.

Conventional biventricular CRT based on right ventricular (RV) and LV pacing is also limited in its ability to fully restore physiological LV activation. Limitations of biventricular CRT may also include the potential desynchronizing effect of RV pacing , non-physiological epicardial LV pacing, latency and suboptimal position of LV lead (paraseptal or apical) due to anatomical features of the target vein, and the presence of LV myocardial scar. The inability of biventricular CRT to restore physiological activation may be expressed in QRS complex widening, rather than in its narrowing. That is observed in a third of patients with biventricular CRT and associated with a poor prognosis.

The combination of LBB and LV pacing may overcome some of the aforementioned limitations of both methods, providing a narrower QRS complex and more effective CRT, especially in difficult cases and in patients with more severe HF. Several studies have shown that combined CRT with LBB and LV pacing is feasible and safe and provides greater electrical resynchronization compared to biventricular CRT.

The above studies demonstrate that LBBP is clinically feasible in patients with HF and LBBB. However, there are still few data about CRT using LBBP in patients with HF and reduced LVEF. There are also only few studies on direct comparison of changes in clinical, speckle tracking echocardiography and other laboratory and instrumental parameters between patients with conventional biventricular CRT and CRT with LBBP.

CRT induces reverse remodeling of the affected heart, improves LV systolic and diastolic function and left heart filling pressure. The measurement of fibrosis and remodeling biomarkers representing the pattern of active processes in HF may be useful.

The relationship between changes in the biomarkers level and reverse remodeling process in patients with LBBP is currently poorly understood. And there are no publications regarding the correlation of the level of such biomarkers as mid-regional pro atrial natriuretic peptide (MR-proANP), growth differentiation factor (GDF)-15, galectin-3, suppression of tumorigenicity 2 (ST2), mid-regional pro adrenomedullin (MR-proADM) and aminoterminal propeptide of type I procollagen (PINP) with clinical and instrumental indicators of patients with LBBP in the available literature. This creates all the prerequisites for studying the association of the above biomarkers with the reverse remodeling process in patients with CRT using LBBP.

ELIGIBILITY:
Inclusion criteria:

1. The patient is willing and able to comply with the protocol and has provided written informed consent;
2. Male or female patients aged 18 to 80 years;
3. Patients with ischemic or non-ischemic cardiomyopathy;
4. Symptomatic HF for at least 3 months prior to enrollment in the study;
5. New York Heart Association (NYHA) functional class HF ≥ II;
6. Patients who are non-responders to biventricular CRT with HF, reduced LVEF and CRT-D replacement or one of the CRT-D leads replacement indications (without LVEF increase ≥ 5% and/or without a left ventricle end-systolic volume decrease ≥ 15% after CRT-D implantation at least 1 year old);
7. Optimal HF medical therapy.

Exclusion criteria:

1. Coronary artery (CA) bypass grafting, balloon dilatation or CA stenting within 3 months prior to enrollment;
2. Acute myocardial infarction within 3 months prior to enrollment;
3. Acute coronary syndrome;
4. Patients with planned cardiovascular intervention (CA bypass grafting, balloon dilatation or CA stenting);
5. Patients listed for heart transplant;
6. Patients with implanted cardiac assist device;
7. Acute myocarditis;
8. Infiltrative myocardial disease;
9. Hypertrophic cardiomyopathy;
10. Severe primary stenosis or regurgitation of the mitral, tricuspid and aortic valves;
11. Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertility age;
12. Mental or physical inability to participate in the study;
13. Patients unable or unwilling to cooperate within the study protocol;
14. Patients with rheumatic heart disease;
15. Mechanic tricuspid valve patients;
16. Patients with any serious medical condition that could interfere with this study;
17. Enrollment in another investigational drug or device study;
18. Patients not available for follow-up;
19. Patients with severe chronic kidney disease (estimated glomerular filtration rate ˂ 30 ml/min/1.73 m2);
20. Life expectancy ≤ 12 months;
21. Participation in another telemonitoring concept.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or worsening of heart failure requiring unplanned hospitalization (%) | 24 month
  Definition of all-cause mortality All deaths and all heart transplants due to the terminal heart failure. Heart transplanted patients will be dropped out and followed in respect of their vital status for the duration of the study.
  Definition of worsening of heart failure requiring unplanned hospitalization Patients requiring intra-venous medication for heart failure (including diuretics, vasodilators or inotropic agents) or a substantial increase in oral diuretic therapy for heart failure (i. e. an increase of Furosemide ≥ 40 mg or equivalent, or the addition of a thiazide to a loop diuretic) will be deemed to have worsening of heart failure. Further, rales and/or S3 sound, chest x-ray, worsening of dyspnoea, worsening of peripheral edema and increase of class NYHA will be assessed for determination of worsening of heart failure. Unplanned hospitalization is defined as any in-hospital stay over one date change, and not planned by the Investigator

SECONDARY OUTCOMES:
All-cause Mortality (%) | 24 month
  As defined for primary endpoint: all deaths and all heart transplants because of terminal heart failure.
Cardiovascular Mortality (%) | 24 month
  All deaths due to cardiovascular reasons and all heart transplants because of terminal HF. Deaths due to worsening of HF, acute coronary syndrome, cerebrovascular accidents, or other cardiovascular events will qualify for this secondary endpoint.
Worsening of Heart Failure Requiring Unplanned Hospitalization (%) | 24 month
  As defined for the primary end-point: patients requiring intra-venous medication for HF (including diuretics, vasodilators, or inotropic agents) or a substantial increase in oral diuretic therapy for HF (i. e. an increase of Furosemide ≥ 40 mg or equivalent, or the addition of a thiazide to a loop diuretic) will be deemed to have worsening of HF. Further, rales and/or S3 sound, chest x-ray, worsening of dyspnoea, worsening of peripheral edema, and increase of class NYHA will be assessed for determination of worsening of HF. Unplanned hospitalization is defined as any in-hospital stay over one date change, and not planned by the Investigator.
  Reasons for worsening of HF may include atrial fibrillation, acute coronary syndrome and hypertension.
Unplanned Hospitalization due to Cardiovascular Reason (%) | 24 month
  Any in-hospital stay over one date change due to cardiovascular reason, which includes worsening of HF, acute coronary syndrome, cerebrovascular accidents, or other cardiovascular events, and not planned by the Investigator.
  In case the hospitalization is classified as planned by the Investigator, and the time interval between the decision to hospitalize and the hospitalization is less than 24 hours.
All-cause Hospitalization (%) | 24 month
  Any in-hospital stay over one date change.
Number of Delivered CRT-D Shocks (n) | 24 month
  An CRT-D shock is an electrical treatment consisting of a high voltage capacitor discharge delivered upon detection of VT/VF episode. All implantable cardioverter-defibrillator (ICD) shocks will be collected and classified by the Investigator as successful or non successful in respect to the termination of the tachyarrhythmia.
Time to First CRT-D Shock (days) | 24 month
  It is the time interval between the end of the 12 weeks blanking after baseline and the first shock. The appropriateness of the therapy will be also assessed.
Number of Delivered CRT-D ATPs (n) | 24 month
  An CRT-D antitachycardia pacing therapy (ATP) is an electrical treatment consisting of timed stimuli delivered upon detection of ventricular tachycardia/ventricular fibrillation (VT/VF) episode. All CRT-D ATPs will be collected and classified by the Investigator as successful or non successful in respect to the termination of the tachyarrhythmia.
Time to First CRT-D ATP (days) | 24 month
  It is the time interval between the end of the 12 weeks blanking after baseline and the first ATP therapy.
Number of Device Detected VT/VF Episodes (n) | 24 month
  It is any ventricular tachyarrhythmia which fulfils the programmed detection criteria of the device in order to be classified as tachyarrhythmic ventricular episode. Device detected episodes will be classified by the Investigator as appropriately detected in presence of real tachyarrhythmia, or inappropriately detected in case of other reasons (oversensing, noise, fast ventricular rate due to supraventricular tachycardia).
Left Ventricular Function (LVEF, %) | 24 month
  The measurement of the left ventricular ejection fraction performed by echocardiography using the modified Simpson's rule.
Exercise Tolerance (m) | 24 month
  It is the measurement of the maximal distance that the patient is able to walk within 6 minutes.
Life Quality (MLWHFQ score) | 24 month
  The life quality is the patient's ability to enjoy normal life activities. For patients suffering from HF, improvement of quality of life is one of the most important goals of new treatments, sometimes as important as improved survival.
  Some medical treatments can seriously impair quality of life without providing appreciable benefit, while others greatly enhance it. To evaluate the effect of cardiac resynchronization therapy with left bundle branch pacing on the quality of life of patients, general and heart failure-related quality of life questionnaires, both filled in by each individual patient, will be used. The Minnesota Living with Heart Failure Questionnaire (MLWHFQ, scale from 0 to 5) will be used.
Life Quality (EuroQol 5-dimensional questionnaire score) | 24 month
  The life quality is the patient's ability to enjoy normal life activities. For patients suffering from HF, improvement of quality of life is one of the most important goals of new treatments, sometimes as important as improved survival.
  Some medical treatments can seriously impair quality of life without providing appreciable benefit, while others greatly enhance it. To evaluate the effect of cardiac resynchronization therapy with left bundle branch pacing on the quality of life of patients, general and heart failure-related quality of life questionnaires, both filled in by each individual patient, will be used. The European Quality of Life Questionnaire (EuroQol 5-dimensional questionnaire, scale from 0 to 100) will be used.

OTHER OUTCOMES:
Echocardiography Left Ventricular Volume Improvement (%) | 24 month
  Echocardiographic measurements will be done at baseline, 6, 12, 18 and 24 month follow-up, to evaluate effect of CRT-D implantation on left ventricle (LV) volume. Improvements due to reverse remodelling of the heart will be evaluated by measuring left ventricular end-systolic volume (LVESV), which is supposed to decrease at follow-up.
  Further, LV volume improvement will be calculated using formula: ((A-B)/A) x 100% (A-baseline LVESV; B-follow-up LVESV).
Echocardiography Left Ventricular Ejection Fraction Improvement (%) | 24 month
  Echocardiographic measurements will be done at baseline, 6, 12, 18 and 24 month follow-up, to evaluate effect of CRT-D implantation on left ventricle (LV) contractility function. Improvements due to reverse remodelling of the heart will be evaluated by measuring left ventricular ejection fraction (LVEF), which is supposed to increase at follow-up. Further, LV contractility function improvement will be calculated using formula: ((A-B)/A) x 100% (A-baseline LVEF; B-follow-up LVEF).
NYHA Class | 24 months]
  The NYHA functional classification provides a simple way of classifying the extent of HF. It is based on questions, related to the usual daily activities and symptoms posed to the patients, and it will be determined at enrollment, baseline and at each follow-up visit. In ablated patients an improvement of NYHA class is expected, the analysis of which will help to assess the efficacy of ablation therapy.
Rate of Drug Support Requirements (%) | 24 month
  Beta-blockers, angiotensin-converting enzyme inhibitors, angiotensin II receptor antagonists, aldosterone antagonists, diuretics, and sodium-glucose transporter type 2 inhibitors, antiarrhythmics and diuretics are drugs commonly taken by patients suffering from HF. Those drugs may have the potential to induce arrhythmic events. In patients with left bundle branch pacing (LBBP) CRT-D a reduction in drug consumption is expected, with a consequent reduction of side effects. The evaluation of the drug regimen will help to assess the effectiveness of LBBP.

CONTACTS AND LOCATIONS:
Overall Officials: Tariel A Atabekov, Ph.D., Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences; Roman E Batalov, M.D., Study Director — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Next individual participant data will be shared with other researchers: gender, age, laboratory and instrumental data
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Starting 12 months after publication
Access Criteria: Principal investigator and study director will review requests and criteria for reviewing requests